CLINICAL TRIAL: NCT02066987
Title: The Effects of Two Volitional Interventions to Improve Oral Health Behaviour Among Iranian Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Vice Chancellor for Research, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QUMS-B23
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Oral Health Behavior Change
Keywords: Action planning, Implementation intention

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Implementation intention (Experimental): It may be helpful for you to plan when and where you will brush your teeth each day over the next month. Please write below when, where, and after what activity you will brush your teeth (e.g., at 8.00 a.m. and 9.00 p.m. in the bathroom after eating breakfast/dinner). Because you should brush your teeth twice a day, please make two plans.
  If it is _____ (WHEN) at or in _______ (WHERE) before/after ______ (ACTIVITY), then I will brush my teeth! If it is _____ (WHEN) at or in _______ (WHERE) before/after ______ (ACTIVITY), then I will brush my teeth!
  Interventions: Behavioral: Implementation intention
- Action planning (Experimental): It may be helpful for you to plan when and where you will brush your teeth each day over the next month. Please write below when, where, and after what activity you will brush your teeth (e.g., at 8.00 a.m. and 9.00 p.m. in the bathroom after eating breakfast/dinner). Because you should brush your teeth twice a day, please make two plans.
  I will brush my teeth at ___(WHEN) at or in ____(WHERE) before/after ___ (ACTIVITY).
  I will brush my teeth at ___(WHEN) at or in ____(WHERE) before/after ___ (ACTIVITY).
  Interventions: Behavioral: Action planning
- active control group (Active Comparator): Participants in the active control group will receive an educational pamphlet containing what it is dental brushing, why it is done, and how it is done.
  Interventions: Behavioral: active control group

INTERVENTIONS:
Behavioral: Implementation intention — It may be helpful for you to plan when and where you will brush your teeth each day over the next month. Please write below when, where, and after what activity you will brush your teeth (e.g., at 8.00 a.m. and 9.00 p.m. in the bathroom after eating breakfast/dinner). Because you should brush your teeth twice a day, please make two plans.
  If it is _____ (WHEN) at or in _______ (WHERE) before/after ______ (ACTIVITY), then I will brush my teeth! If it is _____ (WHEN) at or in _______ (WHERE) before/after ______ (ACTIVITY), then I will brush my teeth!
  Arms: Implementation intention
Behavioral: Action planning — It may be helpful for you to plan when and where you will brush your teeth each day over the next month. Please write below when, where, and after what activity you will brush your teeth (e.g., at 8.00 a.m. and 9.00 p.m. in the bathroom after eating breakfast/dinner). Because you should brush your teeth twice a day, please make two plans.
  I will brush my teeth at ___(WHEN) at or in ____(WHERE) before/after ___ (ACTIVITY).
  I will brush my teeth at ___(WHEN) at or in ____(WHERE) before/after ___ (ACTIVITY).
  Arms: Action planning
Behavioral: active control group — Participants in the active control group will receive an educational pamphlet containing what it is dental brushing, why it is done, and how it is done.
  Arms: active control group

SUMMARY:
the present study had two main aims. First, due to the current underconsumption of dental brush adolescents, the investigators should apply a volitional intervention to increase oral health behvaiour in adolescents. Second, the investigators aim to compare the effectiveness of action planning intervention and implementation intention will improve oral health behavior in adolescents.

DETAILED DESCRIPTION:
This is a study to explore the impact of two volitional interventions on brushing intentions , behaviors and clinical characteristics among a sample of adolescent students.

ELIGIBILITY:
Inclusion Criteria:

* 14 Years to 19 Years
* Ability to understand Persian language Adolescents attending high schools in Qazvin

Exclusion Criteria:

* participate in any kind of oral health education and promotion programs
* undergoing orthodontic treatment

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1110 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
changes in frequencies of dental brushing | changes from baseline, one month after the intervention and six months follow-up

SECONDARY OUTCOMES:
changes in psychological predictors of dental brushing (intention ,perceived behavioural control and Self-monitoring) | changes from baseline, one month after the intervention and six months follow-up
Changes in Community Periodontal Index (CPI) | changes from baseline, one month after the intervention and six months follow-up
Changes in Turesky Modification of the Quigley-Hein Plaque Index | changes from baseline, one month after the intervention and six months follow-up
Oral health related quality of life | changes from baseline and six months follow-up
The frequency of the use of planning | changes from baseline, one month after the intervention and six months follow-up
  The number of planning strategies is used by the adolescents before, at baseline, one month after the intervention and six months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health, Qazvin University of Medical Sciences, Qazvin, Qazvin Province, Iran

REFERENCES:
- [Derived] Pakpour AH, Gholami M, Gellert P, Yekaninejad MS, Dombrowski SU, Webb TL. The Effects of Two Planning Interventions on the Oral Health Behavior of Iranian Adolescents: A Cluster Randomized Controlled Trial. Ann Behav Med. 2016 Jun;50(3):409-18. doi: 10.1007/s12160-015-9767-3. PMID 26791023